CLINICAL TRIAL: NCT03786575
Title: Clinical Value of Next Generation Sequencing in Endocrine Therapy for Advanced Hormone Receptor Positive/HER-2 Negative Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Fei Ma, Deputy Director of Oncology Medicine, Peking Union Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC1787
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2018-11

CONDITIONS: Breast Neoplasm Female; Therapeutics; Mutation
Keywords: Breast Neoplasm; Next Generation Sequencing; Endocrine Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- NGS detection group (Experimental): Before treatment, the patients in the study group underwent NGS detection of ctDNA and formulated endocrine treatment plan according to the test results. After 2 months of endocrine therapy, all patients underwent NGS detection of ctDNA, and the efficacy was evaluated according to RECIST v1.1 standard.
  Interventions: Diagnostic Test: Next Generation Sequencing (NGS) detection

INTERVENTIONS:
Diagnostic Test: Next Generation Sequencing (NGS) detection — The NGS detection panel is designed by our team and covers genes that are clinically useful and have definite guiding significance for endocrine therapy

SUMMARY:
To determine the landscape of gene mutation before and after endocrine therapy, to search for molecular markers of endocrine therapy efficacy, and to explore the clinical value of using NGS detection of ctDNA to guide precise endocrine therapy in patients with advanced breast cancer. The primary endpoints were progression-free survival (PFS), and the secondary endpoints included overall survival time (OS), adverse events (AE), and severe adverse events (SAE).

DETAILED DESCRIPTION:
Before treatment, the patients in the study group underwent NGS detection of ctDNA and formulated treatment plan according to the test results: 1) those with ESR1 mutation and who did not use fulvestrant before, preferred fulvestrant; 2) those with abnormal activation of PI3K/Akt/mTOR pathway signal, preferred mTOR inhibitor combined with endocrine therapy; 3) those with HER-2 sensitive point mutation, preferred anti-HER-2 therapy combined with endocrine therapy; 4) PDGFR mutation, preferential use of PDGFR inhibitors combined with endocrine therapy; 5) no significant gene mutation, making endocrine therapy plan according to the actual clinical situation. After 2 months of endocrine therapy, all patients underwent NGS detection of ctDNA, and the efficacy was evaluated according to RECIST v1.1 standard. If the efficacy evaluation is effective, continue the current treatment and re-evaluate the efficacy every two months; if the efficacy evaluation is ineffective (progress), then withdraw from this study. The vital signs, blood routine, liver and kidney functions and imaging examinations were examined at least every two months in the patients in the study group, and the curative effect was evaluated according to RECIST v1.1 standard.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, female；
2. Pathologically and immunohistochemically confirmed ER-positive/HER-2-negative patients with advanced breast cancer；
3. According to RECIST standard, lesions can be measured (primary lesion length > 1.0 cm or lymph node diameter > 1.5 cm)；
4. Previous endocrine therapy resistance, preparation for second-or-above-line endocrine therapy；
5. No visceral crisis；
6. ECOG PS score: 0-2 points;
7. Laboratory criteria:

   ① white blood cells were more than 4 x 109 /L, and neutrophil count (ANC) was more than 1.5 x 109 /L.

   ② platelet (>100 *109/L); hemoglobin (>10g/dL); serum creatinine (<1.5 *normal value) upper limit (ULN); aspartate aminotransferase (AST) (<2.5 *ULN); alanine aminotransferase (ALT) (<2.5 *ULN); total bilirubin (<1.5 *ULN); serum creatinine (<1.5 *ULN);
8. the volunteers voluntarily joined the study, signed informed consent, and had good compliance and follow-up.

Exclusion Criteria:

1. Pregnant or lactation woman
2. With mental disease
3. With severe infection or active gastrointestinal ulcers
4. With severe liver disease (such as cirrhosis), kidney disease, respiratory disease or diabetes
5. taking part or participating in other clinical trials within one month.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 36 months
  From date of first use endocrine treatment until the date of first documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
Overall survival (OS) | up to 60 months
  Time from first use endocrine treatment to death
Adverse events (AEs) | up to 36 months
  Adverse events (AEs) and laboratory tests graded according to the NCI CTCAE (version 4.0)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided